CLINICAL TRIAL: NCT03404349
Title: Gender-specific Effect of a Tailored, Adolescent Developed Mindfulness Intervention
Brief Title: Tailored Mindfulness Intervention in Adolescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kristen Rawlett, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HP-00077414
Record Dates: First submitted 2017-12-18; First posted 2018-01-19 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Stress; Mindfulness; Affect
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness for Adolescence Course (Experimental): Participants will attend mindfulness classes to include deep breathing, yoga, listening to music and meditation.
  Interventions: Behavioral: Mindfulness for Adolescence Course

INTERVENTIONS:
Behavioral: Mindfulness for Adolescence Course — There are 6 topics that will each be presented over 2 weeks for the 12 week intervention. Individuals will participate in a one to 1.5 hours, once a week intervention for 12weeks. Mindfulness is the practice of becoming aware of one's present-moment experience with compassion and openness as a basis for wise action. This curriculum is intended to strengthen attention and emotion regulation, cultivate wholesome emotions like gratitude and compassion, expand the repertoire of stress management skills, and help participants integrate mindfulness into daily life. Each lesson includes age-appropriate discussion, activities, and opportunities to practice mindfulness in a group setting.

SUMMARY:
Approximately 13%-20% of children living in the United States experience a mental health problem in any given year. Youth with mental illness have difficulty in social settings and have poor academic performance that place them at risk for increased stress and poor mental health outcomes. Stress typically manifests as depression, anxiety, or behavioral issues that lead to increasingly complex treatment with psychotropic medication. It would follow that reducing stress may be a way to improve psychological well being, prevent poor mental health outcomes, and hopefully avoid the need for psychotropic medication. Mindfulness teaching is a potentially powerful tool for adolescents because it focuses on reducing stress. Thus far, studies have not engaged adolescents in developing a patient-centered approach to mindfulness Interventions. The current project would be a significant contribution to clinical practice and the scientific evidence for mindfulness interventions. This research targets psychological well-being within a vulnerable adolescent population that is generally underrepresented in research. The research outcomes will be useful to healthcare providers, educators, and parents/families in encouraging optimal outcomes for adolescents. The overall goals of this proposed research project are to develop and assess the feasibility of an adolescent-developed mindfulness intervention.

DETAILED DESCRIPTION:
At-risk behaviors are related to poor outcomes among adolescents. Increasing evidence supports adolescence as a vital time to introduce stress reduction techniques to reduce risk and improve mental health. The proposed study will develop and test a mindfulness intervention for adolescents in a quasi-experimental pre-test, post-test design.

Mindfulness teaching is a potentially powerful tool for adolescents because it focuses on reducing stress, which can manifest as depression, anxiety or behavioral problems that often are managed with complex psychotropic medication regimens. Thus far, studies have not engaged adolescents in developing mindfulness interventions. Such interventions are critical given that in the United States, 13%-20% of children experience a mental health problem in any given year. Moreover, youth with a mental illness have difficulty in social settings and have poor academic performance that place them at risk for increased stress and poor mental health outcomes. It would follow that reducing stress may be a way to improve psychological well-being, prevent poor mental health outcomes, and hopefully avoid the need for complex psychotropic medication. The overall goals of this proposed research are to develop and to assess the feasibility of an adolescent-developed mindfulness intervention.

The proposed pilot will build from the PI's prior and current research. Earlier research determined that a mindfulness curriculum can have a notable positive impact on affect, coping, and mindfulness in at-risk adolescent girls. This work was expanded by engaging the perspectives of adolescents' from Southwest Baltimore in planning a mindfulness intervention. Earlier research was funded by a pilot grant through an Agency for Healthcare Research and Quality (AHRQ) R24 infrastructure grant to promote patient- centered outcomes research (PCOR) at the University of Maryland Baltimore. The preliminary data for the current proposal is based on these prior studies. The current proposed study, conducted under the Dean's Research Scholar program, will test the impact of a mindfulness intervention on decreasing stress and increasing well-being in adolescents. The specific aims of the pilot study are to:

1. To develop a tailored mindfulness program for adolescents in Southwest Baltimore.
2. To pilot implementation of a tailored a mindfulness program for adolescents residing in Southwest Baltimore.

The proposed study will develop and test a mindfulness intervention for adolescents in a non-randomized convenience sampling, quasi-experimental pre-test, post-test design.Recruitment will occur among middle school students attending public school in Southwest Baltimore. After informed consent and assent, participants will attend mindfulness classes (MC) once per week for 12 weeks. The class content will come from previous pilot work and focus groups, both conducted by the researcher. MC classes will be led by the Holistic Life Foundation. Baseline evaluation will analyze demographics, coping (Response to Stress Questionnaire, RSQ), positive affect (10 item Positive and Negative Affect Scale for Children, PANAS-C) and mindfulness (Mindfulness Attention Awareness Scale, MAAS). In addition, possible gender differences in outcomes will be analyzed. Participants will be contacted 3 months after study completion and again 1 year after study completion to re-evaluate study outcomes via self-reported tools used earlier in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Student at Pinderhughes Middle School
2. In 6-8 grade
3. Parent or legal guardian, confirmed by school records, is 18 years or older
4. Ages 11-13 years old at time of enrollment

Exclusion Criteria:

1. Lack of English fluency in participant or parent/guardian
2. Inability to complete measurement tools
3. Inability to attend the intervention meetings due to school or personal conflicts
4. self-reported pregnancy
5. No wards of the state or emancipated minors

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Response to Stress Questionnaire at 12 weeks, 6 months & 1 year. | 12 weeks, 6 months, 1 year
  Self-Reported primary & secondary coping: The 57-item RSQ instrument was used to evaluate voluntary and involuntary reactions to stressors and was formulated according to varied responses specific to children and adolescents. The measure uses a 4-point Likert response scale (1= No stress or problem coping to 4= A lot of stress or problem coping). Higher scores represent increased use of coping mechanisms. It is recommended that the total score for primary coping be calculated and divided by the total RSQ score to control for response bias and individual differences in base-rates of item endorsement.

SECONDARY OUTCOMES:
Change from Baseline Positive and Negative Affect Schedule for Children at 12 weeks, 6 months & 1 year | 12 weeks, 6 months, 1 year
  Self-reported positive and negative emotions such as happy, joyful, sad & angry: The 10-item PANAS-C was used to measure positive affect (PA).
  The shortened tool was adapted from the 20-item PANAS-C (Laurent et al, 1999). The 10-item PANAS-C provides information regarding affect and can be used in the school or clinic setting. The PA questions (M=16.9, SD=5.5) focus on joyful, cheerful, happy, lively and proud. The measure uses a 5-point Likert response scale (1= Very Slightly or Not at All to 5= Extremely) and the range for each scale is 5-25. The newly formulated 10-item tool shows good reliability and validity with higher scores representing higher levels of positive affect.

OTHER OUTCOMES:
Change from Baseline Mindful Attention Awareness Scale at 12 weeks, 6 months & 1 year | 12 weeks, 6 months, 1 year
  Self-reported state mindfulness: . It places a focus on present time attention and awareness, leaving out dimensions of mindfulness, such as non-judgmental accepting. Statements characterize ideas or actions that are not congruent with mindfulness such as being on automatic pilot, preoccupation and being distracted.
  The 15-item measure uses a 6-point Likert response scale (1= Almost Always to 6= Almost Never) and higher scores indicate higher levels of mindfulness with a possible range of 15-90. Specifically, MAAS demonstrated excellent reliability (-.82- .87) and was validated with multiple studies that demonstrate validity as the correlation between the MAAS and an alternate scale was .70.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinderhughes School, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No